CLINICAL TRIAL: NCT04277520
Title: Postoperative Pain Assessment After Using Different Kinematics During Endodontic Instrumentation (Randomized Clinical Trial)
Brief Title: Postoperative Pain Assessment After Using Different Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Mokhtar Nagy, Associate professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASFD-ENDO-1
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Root Canal Therapy
MeSH Terms: interventions — Root Canal Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continous rotation (Active Comparator): instrumentation was done in continuous rotation motion
  Interventions: Procedure: Root canal therapy
- Reciprocation (Active Comparator): instrumentation was done in reciprocation motion
  Interventions: Procedure: Root canal therapy
- Adaptive motion (Active Comparator): instrumentation was done in adaptive motion
  Interventions: Procedure: Root canal therapy

INTERVENTIONS:
Procedure: Root canal therapy — Different types of instrumentation motions during root canal therapy

SUMMARY:
The aim of this study is to evaluate postoperative pain after endodontic instrumentation using rotation, reciprocation and adaptive motion.

DETAILED DESCRIPTION:
Post operative pain assessment is done at the end of the session Visual Analog Scale (VAS) questionnaires were handed out to the patients and they were asked to assign a number correlating to their post-treatment pain, with 0 representing no pain and 10 representing the most severe pain imaginable.These scores were marked in intervals of 6, 12, 24, 48 and 72 h following endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients with good health.
2. Patient's age between 18_50
3. Mandibular first molars teeth diagnosed clinically and radiographically as acute irreversible pulpitis with no evidence of apical pathosis
4. Positive patient's acceptance for participation in the study

Exclusion Criteria:

* Root resorption
* Non restorable teeth.
* Pregnancy.
* Systematic disease as hypertension ,diabetes .
* Psychologically disturbance.
* Need for prophylactic antibiotics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
monitoring the change in postoperative pain following root canal treatment | 72 hours
  At the end of the session Visual Analog Scale (VAS) questionnaires were handed out to the patients and they were asked to assign a number correlating to their post-treatment pain, following endodontic treatment with 0 representing no pain and 10 representing the most severe pain

SECONDARY OUTCOMES:
6-hour post operative pain assessment | 6 hours
  At the end of the session Visual Analog Scale (VAS) questionnaires were handed out to the patients and they were asked to assign a number correlating to their post-treatment pain after 6 hours, following endodontic treatment with 0 representing no pain and 10 representing the most severe pain
12-hour post operative pain assessment | 12 hours
  At the end of the session Visual Analog Scale (VAS) questionnaires were handed out to the patients and they were asked to assign a number correlating to their post-treatment pain after 12 hours, following endodontic treatment with 0 representing no pain and 10 representing the most severe pain
24-hour post operative pain assessment | 24 hours
  At the end of the session Visual Analog Scale (VAS) questionnaires were handed out to the patients and they were asked to assign a number correlating to their post-treatment pain after 24 hours, following endodontic treatment with 0 representing no pain and 10 representing the most severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hashem, PhD, Study Director — Faculty of Dentistry, Ain Shams university
Locations (1):
- Faculty of Dentistry, Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gambarini G, Testarelli L, De Luca M, Milana V, Plotino G, Grande NM, Rubini AG, Al Sudani D, Sannino G. The influence of three different instrumentation techniques on the incidence of postoperative pain after endodontic treatment. Ann Stomatol (Roma). 2013 Mar 20;4(1):152-5. doi: 10.11138/ads.0152. Print 2013 Jan. PMID 23741536